CLINICAL TRIAL: NCT06307431
Title: A Phase 2, Randomized, Double-blind, Clinical Study of V940 (mRNA-4157) Plus Pembrolizumab (MK-3475) Versus Placebo Plus Pembrolizumab in the Adjuvant Treatment of Participants With Renal Cell Carcinoma (INTerpath-004).
Brief Title: A Study of Adjuvant Intismeran Autogene (V940) and Pembrolizumab in Renal Cell Carcinoma (V940-004).
Acronym: INTerpath-004
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V940-004; 2023-505177-32-00 (Registry Identifier: EU CT); U1111-1291-1851 (Registry Identifier: UTN); V940-004 (Other: MSD)
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intismeran autogene + Pembrolizumab (Experimental): Participants will receive intismeran autogene 1 mg via intramuscular (IM) injection every 3 weeks (Q3W) for up to 9 doses plus Pembrolizumab 400 mg via an intravenous (IV) infusion every 6 weeks (Q6W) for 9 cycles (up to ~54 weeks). Each cycle is 6 weeks.
  Interventions: Biological: Intismeran autogene; Biological: Pembrolizumab
- Placebo + Pembrolizumab (Active Comparator): Participants will receive placebo as an IM injection Q3W for up to 9 doses plus Pembrolizumab 400 mg via an IV infusion Q6W for 9 cycles (up to ~54 weeks). Each cycle is 6 weeks.
  Interventions: Biological: Pembrolizumab; Biological: Placebo

INTERVENTIONS:
Biological: Intismeran autogene — IM injection
  Other Names: mRNA-4157; V940
  Arms: Intismeran autogene + Pembrolizumab
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Biological: Placebo — IM injection
  Arms: Placebo + Pembrolizumab

SUMMARY:
The primary objective of the study is to compare intismeran autogene plus pembrolizumab to placebo plus pembrolizumab in participants with renal cell carcinoma (RCC) with respect to disease-free survival (DFS) as assessed by the investigator. The primary hypothesis is that intismeran autogene plus pembrolizumab is superior to placebo plus pembrolizumab with respect to DFS.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of renal cell carcinoma (RCC) with clear cell or papillary histology.
* Has intermediate-high-risk, high-risk, or M1 no evidence of disease (NED) RCC as defined by the following pathological tumor-node metastasis and tumor grading:
* Intermediate-high-risk RCC: pT2 Gr4, N0, M0; pT3 Gr3/4, N0, M0
* High-risk RCC: pT4, N0, M0; pT any stage, N1, M0
* M1 NED RCC participants who present not only with the primary kidney tumor, but also solid, isolated, soft tissue metastases that can be completely resected at 1 of the following: the time of nephrectomy (synchronous), or ≤2 years from nephrectomy (metachronous)
* Has undergone complete resection of the primary tumor (partial or radical nephrectomy) and complete resection of solid, isolated, soft tissue metastatic lesion(s) in M1 NED participants.
* Must have undergone a nephrectomy and/or metastasectomy ≤12 weeks prior to randomization and recovered from surgery and any post-operative complications before randomization.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before randomization.

Exclusion Criteria:

* Has had a major surgery other than nephrectomy plus resection of preexisting metastases for M1 NED participants, within 4 weeks prior to randomization.
* Has residual thrombus post nephrectomy in the vena renalis or vena cava.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Received prior treatment with a cancer vaccine.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has a history of brain or bone metastatic lesions.
* Has severe hypersensitivity to study medication or any of the substances used to prepare the study medication.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* History of allogeneic tissue/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-01-08 (Estimated); Study Completion 2032-06-08 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | up to ~43 months
  DFS, as assessed by the investigator, is defined as the time from randomization to the first documented local recurrence, or occurrence of distant kidney cancer metastasis(es), or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to ~96 months
  OS is defined as the time from randomization to death due to any cause.
Distant Metastasis-free survival (DMFS) | up to ~ 43 months
  DMFS is defined as the time from randomization to the first diagnosis of a distant metastasis, or death due to any cause, whichever occurs first. Distant metastasis refers to cancer that has spread from the original (primary) tumor to distant organs or distant lymph nodes.
Percentage of Participants Who Experience an Adverse Event (AE) | up to ~15 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The percentage of participants that experience at least one AE will be reported.
Percentage of Participants Who Discontinue Study Treatment Due to an AE | up to ~12 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The percentage of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (63):
- United States (11):
  - City of Hope Comprehensive Cancer Center-Medical Oncology ( Site 0104), Duarte, California
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 140)-Department of Urology/Institute of Uro, Los Angeles, California
  - UCSF Medical Center at Mission Bay ( Site 0108), San Francisco, California
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 0102), New Haven, Connecticut
  - Beth Israel Deaconess Medical Center-Cancer Clinical Trials Office ( Site 0109), Boston, Massachusetts
  - Dana-Farber Cancer Institute-GU ( Site 0101), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center ( Site 0100), New York, New York
  - Duke Cancer Institute ( Site 0106), Durham, North Carolina
  - Abramson Cancer Center ( Site 0107), Philadelphia, Pennsylvania
  - Fox Chase Cancer Center ( Site 0111), Philadelphia, Pennsylvania
  - UT Southwestern Medical Center ( Site 0110), Dallas, Texas
- Argentina (5):
  - Hospital Británico de Buenos Aires-Oncology ( Site 1106), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming-Alexander Fleming ( Site 1101), Buenos Aires, Buenos Aires F.D.
  - Asociación de Beneficencia Hospital Sirio Libanés ( Site 1110), Buenos Aires, Buenos Aires F.D.
  - Centro Privado de RMI Rio Cuarto ( Site 1104), Río Cuarto, Córdoba Province
  - Fundacion Estudios Clinicos ( Site 1111), Rosario, Santa Fe Province
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 1502), Macquarie University, New South Wales
  - Westmead Hospital ( Site 1501), Westmead, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Si, Brisbane, Queensland
  - Fiona Stanley Hospital-Medical Oncology ( Site 1503), Murdoch, Western Australia
- Canada (2):
  - BC Cancer Vancouver ( Site 0005), Vancouver, British Columbia
  - CHU de Quebec - Université Laval - Hotel Dieu de Quebec ( Site 0008), Québec, Quebec
- Chile (4):
  - FALP-UIDO ( Site 1202), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Centro del Cáncer ( Site 1205), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 1201), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS-ACEREY ( Site 1200), Viña del Mar, Región de Valparaíso
- France (5):
  - CENTRE LEON BERARD ( Site 0305), Lyon Cedex08, Auvergne-Rhône-Alpes
  - CHU Besançon ( Site 0302), Besançon, Doubs
  - Institut Claudius Regaud ( Site 0303), Toulouse, Haute-Garonne
  - Hôpital Européen Georges Pompidou ( Site 0300), Paris
  - Gustave Roussy ( Site 0304), Villejuif, Île-de-France Region
- Germany (6):
  - Klinikum Stuttgart - Katharinenhospital ( Site 0400), Stuttgart, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen-Urologische Klinik und Poliklinik ( Sit, Munich, Bavaria
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Urologie ( Site 0405), Dresden, Saxony
  - Universitätsklinikum Jena ( Site 0402), Jena, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0401), Berlin
  - Asklepios Altona-Department of Urology ( Site 0410), Hamburg
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 0501), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0500), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 0504), Florence, Tuscany
  - Azienda Ospedaliero Universitaria di Parma ( Site 0503), Parma
- Poland (3):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 0701), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Moczowego ( S, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0702), Koszalin, West Pomeranian Voivodeship
- South Korea (4):
  - Seoul National University Hospital ( Site 1600), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 1603), Seoul
  - Asan Medical Center ( Site 1602), Seoul
  - Samsung Medical Center ( Site 1601), Seoul
- Spain (3):
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 0801), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0800), Barcelona
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 0802), Seville
- Taiwan (4):
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 1701), Kaohsiung Niao Sung Dist, Kaohsiung
  - China Medical University Hospital-Department of Urology ( Site 1702), Taichung
  - Taichung Veterans General Hospital ( Site 1704), Taichung
  - Taipei Veterans General Hospital ( Site 1703), Taipei
- Turkey (Türkiye) (3):
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 0901), Ankara
  - Ankara Universitesi Tip Fakultesi Hastanesi-Oncology ( Site 0902), Ankara
  - Ege Universitesi Hastanesi-Medical Oncology ( Site 0903), Izmir
- United Kingdom (5):
  - Addenbrooke's Hospital ( Site 1004), Cambridge, Cambridgeshire
  - Gartnavel General Hospital-Clinical Trials Unit ( Site 1002), Glasgow, Glasgow City
  - St Bartholomew's Hospital ( Site 1000), London, London, City of
  - Western General Hospital ( Site 1003), Edinburgh, Midlothian
  - The Christie NHS Foundation Trust ( Site 1001), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26312&tenant=MT_MSD_9011